CLINICAL TRIAL: NCT05705414
Title: Oral Intradialytic Amino Acids Supplementation to Vitalize End-stage Kidney Disease Patients on Hemodialysis (OASIS)
Brief Title: Oral Intradialytic Amino Acid Supplementation to Vitalize End-stage Kidney Disease Patients on Hemodialysis
Acronym: OASIS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); IIMS-UT Health San Antonio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSC20220558H; KL2TR002646 (NIH)
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: End Stage Renal Disease
Keywords: Fatigue; End-stage kidney disease; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Fatigue | interventions — Valine

STUDY DESIGN:
Intervention Model Description: The study design will consist of a crossover schema, with one arm starting on amino acid Valine and the other on EAA for a period of 8 weeks, followed by a washout period of 1 week, and then assignment to the nutritional supplement that they have not already taken for the remaining 8 week period that they are participating in this study.
Masking Description: The intervention will be administered to the subjects by appropriately trained delegates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment group Valine then EEA (Experimental): Valine will be administered as two 4 gm packets administered on dialysis treatment day followed by a washout period and then EEA
  Interventions: Drug: Valine; Drug: EEA
- Treatment group EEA then Valine (Experimental): EAA will be administered as one 12.5 gm packet administered on dialysis treatment day followed by a washout and then Valine
  Interventions: Drug: Valine; Drug: EEA

INTERVENTIONS:
Drug: Valine — A medical food intended for use under medical supervision
  Other Names: Valine Amino Acid Supplement
Drug: EEA — A medical food intended for use under medical supervision
  Other Names: Essential Amino Acid Supplement

SUMMARY:
The study will test and compare the efficacy of a single essential amino acid valine with a combination of essential amino acids (EAA) supplement on fatigue, frailty, and cognitive function in end-stage kidney disease (ESKD) patients undergoing hemodialysis (HD) treatment.

DETAILED DESCRIPTION:
This single center outpatient study will test and compare the efficacy of a single essential amino acid, valine with a combination of essential amino acids (EAA) supplementation on fatigue, fragility and cognitive function in end-stage kidney disease (ESKD) patients aged 18-64 years undergoing hemodialysis (HD) treatment at least three times a week.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age 18-64 years
3. Receiving 3 x weekly in clinic hemodialysis for at least 6 months

Exclusion Criteria:

1. Hypersensitivity to amino acid(s) and/or any excipient
2. Clinical documentation of COVID-19
3. Concomitant intake of amino acids supplements
4. Current use or abuse of alcohol, marijuana, narcotic, or other substances
5. Heart failure receiving active management
6. Malignant cancer receiving anticancer therapy
7. Diagnosis of major depressive disorder receiving antidepressants
8. Diagnosis of chronic liver disease
9. Cerebrovascular disease with sequelae
10. Upper limb amputation, osteoarthritis, or degenerative diseases of fingers, carpel tunnel syndrome in the non-fistula or graft hand preventing completion of hand grip strength test.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Brief Fatigue Inventory (BFI) score | Baseline to 17 weeks
  Changes in global fatigue score measured with the 9-item Brief Fatigue Inventory (BFI). The first 3 questions assess fatigue severity, and the remaining 6 questions measure the impact of fatigue on activity, mood, walking, work, relationships, and enjoyment of life. Respondents rate each item on a 0-10 numeric scale, with 0 meaning "no fatigue" and 10 meaning "fatigue as bad as you can imagine." Scores of all 9 items yield global fatigue burden. A lower average global fatigue score indicates milder fatigue and a higher score severe fatigue.

SECONDARY OUTCOMES:
Handgrip strength test | Baseline to 17 weeks
  Change in handgrip strength measured by a dynamometer in lbs
Trail Making Test (TMT) | Baseline to 17 weeks
  Change in minutes to complete Trail Making Test (TMT) A and B

OTHER OUTCOMES:
Dialysate level of amino acids | Baseline to 17 weeks
  How is this measured, are there different values for different aa's (if so each one should be reported separately)?
Plasma level of amino acids | Baseline to 17 weeks
  How is this measured, are there different values for different aa's (if so each one should be reported separately)?
Blood valine metabolite 3-hydroxyisobutyrate (3-HIB) | Baseline to 17 weeks
  Change in 3-hydroxyisobutyrate (3-HIB) levels
Blood valine beta-amino-isobutyric acid (BAIBA) | Baseline to 17 weeks
  Change in beta-amino-isobutyric acid (BAIBA)

CONTACTS AND LOCATIONS:
Overall Officials: Subrata Debnath, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.
Supporting Information: Study Protocol, SAP
Time Frame: At study completion, once data is published in a peer review journal